CLINICAL TRIAL: NCT00847691
Title: GENSARC 2008 : Medical Economic Evaluation of the Molecular Detection by FISH (Fluorescent in Situ Hybridization) and by PCR (Polymerase Chain Reaction) of Sarcomas Specific Translocations and Amplifications .
Acronym: GENSARC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PSTIC GENSARC
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2009-02

CONDITIONS: Sarcoma
Keywords: economic evaluation; diagnostics; sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — sarcoma biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sarcoma: patients with biopsy or excision of sarcoma (suspected or diagnosed)

SUMMARY:
The clinical and histological diagnosis of sarcomas is often very difficult. The identification of chromosomal and molecular anomalies, such as amplifications, deletions or fusion genes is a powerful help for establishing a correct diagnosis of sarcomas and their benign counterparts. However, the cost of the cytogenetic and molecular techniques for the detection of these alterations is often a limitation to their use. The aim of our study is to evaluate the direct cost of the molecular techniques in comparison to the cost that would be generated by an appropriate therapy and care management of the patient in case of an erroneous diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with biopsy or excision of sarcoma (suspected or diagnosed)
* sampling reviewed by pathologists
* frozen sampling
* clinical data available

Exclusion Criteria:

* opposition of patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a strong clinical and histological suspicion of sarcoma
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence PEDEUTOUR, PhD, Principal Investigator — Laboratoire de Génétique des Tumeurs Solides
Locations (8):
- France (8):
  - Departement de Pathologie de l'Institut Bergonié, Bordeaux
  - Laboratoire de Biochimie et Biologie Moléculaire, CHRU de Lille, Lille
  - Département d'Anantomie et de Cytologie Pathologie, Centre Léon Berard, Lyon
  - Laboratoire de Génétique des Tumeurs Solides, Nice
  - Institut Curie, Paris
  - Service d'Anatomo-Pathologie, Centre Paul Strauss, Strasbourg
  - Unité de Biologie Moléculaire, CHU de Hautepierre, Strasbourg
  - Département de biologie et de pathologie médicales, Institut Gustave roussy, Villejuif